CLINICAL TRIAL: NCT03080805
Title: A Randomised, Open-label, Parallel Controlled, Multicentre, Phase 3 Clinical Trial of Pyrotinib Plus Capecitabine Versus Lapatinib Plus Capecitabine in Patients With HER2+ Metastatic Breast Cancer:
Brief Title: Pyrotinib Plus Capecitabine Versus Lapatinib Plus Capecitabine in Patients With HER2+ Metastatic Breast Cancer. (PHOEBE)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-Ⅲ-MBC
Record Dates: First submitted 2017-03-03; First posted 2017-03-15 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: HER2 Positive Metastatic Breast Cancer
MeSH Terms: interventions — pyrotinib; Capecitabine; Lapatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pyrotinib Plus Capecitabine (Experimental)
  Interventions: Drug: Pyrotinib Plus Capecitabine
- Lapatinib Plus Capecitabine (Active Comparator)
  Interventions: Drug: Lapatinib Plus Capecitabine

INTERVENTIONS:
Drug: Pyrotinib Plus Capecitabine — pyrotinib(400 mg once daily) + capecitabine (2000 mg/m^2 daily, 1000 mg/ m^2 BID)
  Arms: Pyrotinib Plus Capecitabine
Drug: Lapatinib Plus Capecitabine — Lapatinib (1250 mg once daily)+ capecitabine (2000 mg/m^2 daily, 1000 mg/m^2 BID)
  Arms: Lapatinib Plus Capecitabine

SUMMARY:
Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. This study is a randomized,open-label,multi-center,active-controlled, parallel design study of the combination of pyrotinib and capecitabine versus Lapatinib plus capecitabine in HER2+ MBC patients, who have prior received taxane and trastuzumab.Patients will be randomized in a 1:1 ratio to one of the following treatment arms.Arm A: pyrotinib (400 mg once daily) + capecitabine (1000 mg/m^2 twice daily),Arm B: Lapatinib (1250 mg once daily) + capecitabine (1000 mg/m^2 twice daily).Patients will receive either arm of therapy until disease progression, unacceptable toxicity, or withdrawalof consent.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 and ≤70 years.
2. ECOG performance status of 0 to 1.
3. Life expectancy of more than 12 weeks.
4. According to RECIST 1.1, at least one measurable lesion exists
5. Histologically or cytologic confirmed HER2 positive metastatic breast cancer.
6. Prior treatment with trastuzumab (≥2 cycles in metastatic setting, or

   ≥3 months in adjuvant/neoadjuvant setting) and Taxane(≥2 cycles in any setting or untill unendurable AE or progression during treatment).
7. Previously reveived ≤2 chemotherapy regimens in metastasis setting;
8. Required laboratory values including following parameters:

   ANC: ≥ 1.5 x 10^9/L; Platelet count: ≥ 90 x 10^9/L; Hemoglobin: ≥ 90 g/L; Total bilirubin: ≤ 1.5 x upper limit of normal (ULN); ALT and AST: ≤ 2 x ULN(patients with liver metastases: ≤5 x ULN); BUN and Creatinine:

   ≤ 1x ULN;CCR≥50 mL/min;LVEF: ≥ 50%;QTcF: < 450 ms (male)，< 470 ms（female）;
9. Signed informed consent.

Exclusion Criteria:

1. Received capecitabine in metastatic setting;
2. Received HER2 targeted tyrosine kinase inhibitor (including Lapatinib, Neratinib and Pyrotinib);
3. Cumulated dosage of Doxorubincin >400 mg/m^2 or Epirubicin >800 mg/m^2 or equal dosage of other anthracycline drugs in adjuvant/neoadjuvant/metastatic setting );
4. Received surgery，chemotherapy,radiotherapy or target therapy within 28 days prior to randomization. Received hormone therapy within 7 days prior to randomization;
5. Participated in other clinical trial within 28 days prior to randomization.
6. Known dihydro pyrimidine dehydrogenase（DPD）defect;
7. CT or MRI confirmed brain metastases;
8. Bone or skin lesion as unique target lesion;
9. Second malignancies within 5 years, except for cured skin basal cell carcinoma,carcinoma in-situ of uterine cervix and squamous-cell carcinoma;
10. Factors influencing the usage of oral administration (e.g. unable to swallow, chronic diarrhea and intestinal obstruction, etc.);
11. Uncontrolled third space effusion (such as pleural fluid and ascites) by drainage or other clinical intervention;
12. Receiving any other anti-tumour therapy after informed consent;
13. Unprogressed after or during the last anti-tumour therapy,according to RECIST1.1;
14. History of any kind of Heart disease,including 1)Angina pectoris; (2) Arrhythmia required medication or with clinical significance; (3) Myocardial infarction; (4) Heart failure; (5) Any other heart disease judged by researcher as not suitable for participating in this study, etc;
15. History of Immunodeficiency, acquired or congenital immunodeficiency (HIV positive) ,history of organ transplantation;
16. History of neurological or psychiatric disorders, including epilepsy or dementia;
17. Concomitant disease judged by investigators that may bring serious harm to the safety of patients or the completion of this study;
18. All female patients in breastfeeding period or in child-bearing period or with positive pregnancy test result or refusing to take a reliable method of birth control during the study;
19. Any other situations judged by investigator as not suitable for participating in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | Estimated 10 months
  From infromed consent to progression or death

SECONDARY OUTCOMES:
Safety: AE | AE recorded from infromed consent to 28 days after treatment completion
  AE
Overall Survival (OS) | Estimated 30 months
  From infromed consent to death
Objective Response Rate (ORR) | Estimated 10 months
  CR+PR
Time to Progression (TTP) | Estimated 10 months
  From infromed consent to progression
Duration of Response (DOR) | Estimated 10 months
  CR+PR+SD
Clinical Benefit rate (CBR) | Estimated 10 months
  CR+PR+SD≥24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital,Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bao Y, Zhang Z, He X, Cai L, Wang X, Li X. Cost-Effectiveness of Pyrotinib Plus Capecitabine versus Lapatinib Plus Capecitabine for the Treatment of HER2-Positive Metastatic Breast Cancer in China: A Scenario Analysis of Health Insurance Coverage. Curr Oncol. 2022 Aug 23;29(9):6053-6067. doi: 10.3390/curroncol29090476. PMID 36135045
- [Derived] Xu B, Yan M, Ma F, Hu X, Feng J, Ouyang Q, Tong Z, Li H, Zhang Q, Sun T, Wang X, Yin Y, Cheng Y, Li W, Gu Y, Chen Q, Liu J, Cheng J, Geng C, Qin S, Wang S, Lu J, Shen K, Liu Q, Wang X, Wang H, Luo T, Yang J, Wu Y, Yu Z, Zhu X, Chen C, Zou J; PHOEBE Investigators. Pyrotinib plus capecitabine versus lapatinib plus capecitabine for the treatment of HER2-positive metastatic breast cancer (PHOEBE): a multicentre, open-label, randomised, controlled, phase 3 trial. Lancet Oncol. 2021 Mar;22(3):351-360. doi: 10.1016/S1470-2045(20)30702-6. Epub 2021 Feb 11. PMID 33581774